CLINICAL TRIAL: NCT01066403
Title: Dopaminergic Modulation of Prefrontal Functions in Schizophrenic Patients: Adjuvant Therapy With Pergolide
Brief Title: Adjuvant Therapy With Pergolide in Treating Cognitive Deficits in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Daniela Roesch Ely, PI, University of Heidelberg
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 03T-342-DRE
Record Dates: First submitted 2010-02-09; First posted 2010-02-10 (Estimated); Last update posted 2010-02-10 (Estimated); Status verified 2008-12

CONDITIONS: Schizophrenia
Keywords: schizophrenia; cognitive deficits; dopamine; dopamine agonists; prefrontal cortex; D1 specific modulation; pergolide; executive control; working memory; Influence of pergolide on cognition in Schizophrenia; D1-specific modulation of prefrontal functions; Influence of pergolide on psychopathology and depression; Influence of pergolide on extrapyramidal symptoms
MeSH Terms: conditions — Schizophrenia; Cognition Disorders; Depression | interventions — Pergolide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pergolide (Experimental): Patients will be randomly assigned to a sequence of treatments of either pergolide or placebo p.o. under continuous concomitant atypical neuroleptic therapy (stable at least 2 weeks prior trial begin).
  Interventions: Drug: Pergolide

INTERVENTIONS:
Drug: Pergolide — 0,3 mg pergolide (the first two days begin with 0,05mg, then increase of dose of 0,1mg every 3 days for a maximum of 0,3mg/d, taken orally 3x 0,1mg/day). Then stable dose of 0,3mg for one week.. Subsequently slow (for 8 days) reduction of dosage of 0,1mg every 3 days for 6 days then 0,05mg every day for the last two days.
  Placebo group is identical in appearance and number of placebo capsules, in the same starting and maintenance scheme as for the pergolide group.
  Other Names: Parkotil; Pergolid

SUMMARY:
The objective of this study is to compare the modulation of pergolide, a D1/D2 receptor agonist, to placebo in non-acute schizophrenic subjects under concomitant therapy with atypical antipsychotics on specific PFC functions. Further aims are to assess the influence of pergolide on psychopathology and extrapyramidal symptoms in comparison to placebo.

DETAILED DESCRIPTION:
Additionally to the desired treatment of positive symptoms, the administration of typical neuroleptics can lead to undesired side effects such as increase of negative symptomatic and cognitive deficits. The influence of atypical neuroleptics on cognition is still not very well studied. Furthermore there is evidence that some cognitive symptoms seen in schizophrenia are related to a disturbance in the prefrontal cortex PFC and involve specific subtypes of dopamine receptors, namely D1 subtypes, which predominates in this area. It is assumed that patients with this spectrum of cognitive deficits have the worse course and prognosis. Furthermore these deficits are more therapy resistant to the conventional current therapy approaches. There is however some evidence pointing to a positive influence of dopamine agonists on these deficits, but the selective effect of dopamine sub-receptors is still not well investigated. The aim of the study is to examine whether cognitive deficits in higher cognitive functions of the PFC such as working memory, semantic association and executive control improves under dopamine agonistic therapy in schizophrenia and whether this is related to selective D1 modulation.

We predict that the modulation of D1 subtype receptors improve performance in each of these tasks. Because there is no D1 agonist available for human research we decided to use a design comparing a dopamine agonist with mixed D1 and D2 agonistic properties (pergolide) to placebo under a stable D2 antagonistic continuous-therapy with atypical antipsychotics. With this design the D2-component of pergolide can be antagonized by the atypical antipsychotics and a D1 agonistic effect can be suggested, as well as protecting patients against a psychotic re-exacerbation. With this study we aim to bring more insight in the therapy of PFC cognitive deficits of schizophrenia by helping to elucidate the role of selective agonists on cognition in schizophrenic patients. I

ELIGIBILITY:
Inclusion Criteria:

* Non-acute in- and outpatients, with predominantly negative symptoms, and remitted from positive symptoms like hallucinations and delusions for 1 week, with the diagnosis of schizophrenia (ICD 10: F20) at the Psychiatry Hospital of the Universities of Heidelberg, Hamburg-Eppendorf, Zentralinstitut für Seelische Gesundheit Mannheim, SRH Klinikum Karlsbad - Langensteinbach (Clinical interview to establish diagnosis with DSM-IV (M.I.N.I International Neuropsychiatric Interview _ German Version 5.0.0)
* Verbal IQ higher than 80, as measured by the Mehrfachwahl-Wortschatz-Intelligenztest
* Visual acuity must be normal or corrected.
* Color sight intact
* Positive neuroleptics drug monitoring level
* Females must be under adequate contraception (oral hormonal contraceptive, IntraUterineDevice)

Exclusion Criteria:

* Concomitant neurologic and internistic diseases (especially cardiovascular diseases and others like untreated thyroid hyper-/hypofunction, liver or kidney dysfunction, seizures or history of traumatic brain injury)
* Known allergy reaction under ergoline-therapy
* Actual history of drug abuse/addiction, concomitant other psychiatric disorder (screened by SCID) and suicide attempt in the medical history
* Other long term pharmacological treatment which can interact with dopamine agonists and antagonists (e.g. anticoagulants, digitoxin)
* Pregnancy and breastfeeding (anamneses and pregnancy test in urine)
* Participation in other clinical trial for the last 3 months
* History of malignant neuroleptic syndrome

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2003-10; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The D1-specific dopaminergic modulation of prefrontal functions (executive control, working memory, control of semantic association) confirmed by a complex neuropsychological battery including a non - PFC activating control task | 30 days

SECONDARY OUTCOMES:
Influence of pergolide on psychopathology symptoms and extrapyramidal symptoms in comparison to placebo measured by specific rating scales, e.g. PANSS and Calgary Depression Scale | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Roesch - Ely, MD, Principal Investigator — Psychiatrische Universitätsklinik Heidelberg
Locations (4):
- Germany (4):
  - Zentralinstitut für Seelische Gesundheit, Mannheim, 68159
  - Psychiatrische Universitätsklinik, Heidelberg, Baden-Wurttemberg
  - Universitätsklinikum Hamburg - Eppendorf, Hamburg
  - SRH Klinikum Karlsbad - Langensteinbach gGmbH, Karlsbad

REFERENCES:
- See also: Related Info — http://www.klinikum.uni-heidelberg.de/Dopamin-und-Schizophrenie.5472.0.html
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/16721703?ordinalpos=8&itool=EntrezSystem2.PEntrez.Pubmed.Pubmed_ResultsPanel.Pubmed_DefaultReportPanel.Pubmed_RVDocSum